CLINICAL TRIAL: NCT04250519
Title: Assessment of Post Operative Pain Following Root Canal Retreatment in Molars Using Four Different Combination of Irrigants : A Prospective Clinical Study
Brief Title: Evaluation of Post Operative Pain in Retreatment of Molars Using Different Irrigant
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Responsible Party: Principal Investigator, Dr. CT. VALLIAPPAN, Principal Investigator, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TamilNaduMU
Record Dates: First submitted 2020-01-22; First posted 2020-01-31 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Root Canal Infection
MeSH Terms: interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1% sodium hypochlorite & dexamethasone 4mg as irrigants (Experimental): sodium hypochlorite is effective in any concentration as antimicrobial irrigant and dexamethasone is anti inflammatory drug
  Interventions: Drug: Sodium Hypochlorite
- 1% sodium hypochlorite as irrigant &normal saline as placebo (Active Comparator): sodium hypochlorite is effective in any concentration as irrigant
  Interventions: Drug: Sodium Hypochlorite
- 5.25% sodium hypochlorite and dexamethasone 4mg as irrigants (Experimental): sodium hypochlorite is effective in any concentration as antimicrobial irrigant and dexamethasone is anti inflammatory drug
  Interventions: Drug: Sodium Hypochlorite
- 5.25% sodium hypochlorite &normal saline as placebo (Active Comparator): sodium hypochlorite is effective in any concentration as irrigant
  Interventions: Drug: Sodium Hypochlorite

INTERVENTIONS:
Drug: Sodium Hypochlorite — Sodium hypochlorite is used as intracanal irrigant to minimize the post operative pain

SUMMARY:
This study evaluates the efficacy of dexamethasone as a intracanal irrigant along with sodium hypochlorite 1% and 5.25% concentrations in post treatment pain for molar root canal retreatment.

DETAILED DESCRIPTION:
Main objective of root canal retreatment is to alleviate pain and disinfect the rootcanal .However some patients may experience mild to severe pain following treatment , which leads to intake of painkillers orally for post operative pain management.

So , this study evaluates the efficiency of dexamethasone used as intracanal irrigant in post treatment pain for molar root canal retreatment sodium hypochlorite (1% &5.25%) is used for disinfecting the canals patients will be grouped into Symptomatic and Asymptomatic patients requiring root canal retreatment and irrigants will be used in various combinations as mentioned below

1. 1% sodium hypochlorite alone 2.5ml in each canal along with ultrasonic activation
2. 1% sodium hypochlorite and dexamethasone 4mg,2.5ml in each canal along with ultrasonic activation
3. 5.25% sodium hypochlorite alone 2.5ml in each canal along with ultrasonic activation
4. 5.25% sodium hypochlorite and dexamethasone 4mg, 2.5ml in each canal along with ultrasonic activation calcium hydroxide is commonly used as intracanal medicament in all the patients post operative symptoms is evaluated at 12 hrs , 24 hrs,48 hrs, 72 hrs and 1 week followed by obturation is completed

ELIGIBILITY:
Inclusion Criteria:

* teeth previously treated or attempted root canal treatment,
* teeth with or without symptoms,
* periapical radiograph showing evidence of inadequate previous root canal treatment or periapical changes,
* only teeth or at least one canal where complete removal of root canal filling material was possible and reach the working length in first appointment.

Exclusion Criteria:

* patient not willing for follow up,
* teeth with extensive cervical or apical resorption that restricted the use of sodium hypochlorite irrigation,
* teeth with poor periodontal status, teeth not suitable for post endodontic restoration,
* patients with acute periapical abscess,
* patients with systemic conditions preventing radiograph exposure or multi visit treatment,
* pregnant patients,
* patients with allergy to any known dental materials.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
post operative pain evaluation using various combination of irrigants: VAS score | At 6 hours
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .
post operative pain evaluation using various combination of irrigants: VAS score | At 12 hours
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .
post operative pain evaluation using various combination of irrigants: VAS score | At 24 hours
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .
post operative pain evaluation using various combination of irrigants: VAS score | At 48 hours
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .
post operative pain evaluation using various combination of irrigants: VAS score | At 72 hours
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .
post operative pain evaluation using various combination of irrigants: VAS score | After 7 days
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain .

SECONDARY OUTCOMES:
assessment of other variables in pain scale | through study completion, an average of 1 week
  comparing the pain scale experienced between male and female in VAS score
assessment of other variables in pain scale | through study completion, an average of 1 week
  comparing the pain scale experienced between mandibular molar and maxillary molar from VAS score
assessment of other variables in pain scale | through study completion, an average of 1 week
  comparing the pain scale based on patients pre operative symptom ex; patient is symptomatic or Asymptomatic before treatment procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CSI college of dental sciences and research, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: from may 2021 and available till may 2025